CLINICAL TRIAL: NCT01272349
Title: Intermittent Hypoxia Elicits Prolonged Restoration of Motor Function in Human SCI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Shirley Ryan AbilityLab (Other); Shepherd Center, Atlanta GA (Other); Northwestern University (Other); University of Wisconsin, Madison (Other); University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Randy D. Trumbower, Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00035986a; W81XWH-10-1-0832 (Other: Other)
Record Dates: First submitted 2011-01-04; First posted 2011-01-07 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; walking; low oxygen; air; strength
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low oxygen (Experimental)
  Interventions: Other: Acute intermittent hypoxia
- Room Air (Sham Comparator)
  Interventions: Other: Room air

INTERVENTIONS:
Other: Acute intermittent hypoxia — 30 minutes of intermittent breathing low oxygen followed by walking on a body-weight support treadmill
  Other Names: breathing low oxygen
  Arms: Low oxygen
Other: Room air — 30 minutes of breathing room air followed by walking on a body-weight support treadmill
  Other Names: breathing room air
  Arms: Room Air

SUMMARY:
The goal of the study is to determine whether repeatedly breathing low oxygen levels for brief periods (termed intermittent hypoxia) will improve limb function after spinal cord injury. This idea stems from animal studies on respiration, in which investigators have shown that mild intermittent hypoxia improves breathing in spinally injured rats. These studies have shown that intermittent hypoxia induces spinal plasticity, strengthening neural connections and motor neuron function within the spinal cord. Exposure to mild intermittent hypoxia triggers a cascade of events, including increased production of key proteins and increased sensitivity of spinal cord circuitry necessary for improved breathing.

The ultimate goal of this research is to assess the potential of mild intermittent hypoxia as a therapeutic approach to stimulate recovery of limb function in human patients.

DETAILED DESCRIPTION:
: The goal of the study is to determine whether repeatedly breathing low oxygen levels for brief periods (termed intermittent hypoxia) will improve limb function after spinal cord injury. This idea stems from animal studies on respiration, in which investigators have shown that mild intermittent hypoxia improves breathing in spinally injured rats. These studies have shown that intermittent hypoxia induces spinal plasticity, strengthening neural connections and motor neuron function within the spinal cord. Exposure to mild intermittent hypoxia triggers a cascade of events, including increased production of key proteins and increased sensitivity of spinal cord circuitry necessary for improved breathing.

The investigators initially hypothesize that daily exposure to intermittent hypoxia for 7 consecutive days will improve limb function in rats and in humans with chronic spinal injuries. First, the investigators will compare limb function in spinally-injured rats which receive mild intermittent hypoxia treatment with rats that did not. The investigators will measure grip strength and locomotor abilities in both groups before treatment and for several months after treatment. The investigators will also examine the spinal cords of these rats to look for the key proteins, which are indicators of spinal plasticity. The investigators will use this information to guide the treatment protocols when the investigators compare limb function in spinal-injured persons with and without intermittent hypoxia treatment.

The second hypothesis is that combining intermittent hypoxia with locomotor training will further improve limb function after spinal injury. To test this idea, the investigators will compare limb function in spinally-injured rats which have received combined intermittent hypoxia and treadmill training with rats which only received intermittent hypoxia or locomotor training alone. The investigators will examine key proteins in the spinal cords of these rats to determine whether the combination of hypoxia and training further alters these indicators of plasticity. The investigators will also compare limb function in spinally-injured humans who receive both intermittent hypoxia and locomotor treadmill training with those who receive either treatment alone.

The ultimate goal of this research is to assess the potential of mild intermittent hypoxia as a therapeutic approach to stimulate recovery of limb function in human patients.

ELIGIBILITY:
Inclusion Criteria:

* medical clearance to participate
* lesion below C5 and above T12 with non-progressive etiology
* classified as motor-incomplete
* injury greater than 12 months
* ambulatory with minimal assistance

Exclusion Criteria:

* Concurrent severe medical illness (i.e., infection, cardiovascular disease, ossification, recurrent autonomic dysreflexia, unhealed decubiti, and history of cardiac or pulmonary complications)
* Pregnant women because of the unknown affects of AIH on pregnant women and fetus
* History of seizures, brain injury, and/or epilepsy
* Diagnosed with obstructive sleep apnea
* Undergoing concurrent physical therapy
* Any contraindications to EMG testing procedures (skin sensitivity)
* Any contraindications to passive movement of the limbs (e.g., joint immobility, hemodynamic instability)
* Score of < 24 on Mini-Mental Exam

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Walking performance | 1 Week

CONTACTS AND LOCATIONS:
Overall Officials: Randy D Trumbower, PT, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Shepherd Center, Atlanta, Georgia
  - Rehabilitation Institute of Chicago, Chicago, Illinois

REFERENCES:
- [Derived] Hayes HB, Jayaraman A, Herrmann M, Mitchell GS, Rymer WZ, Trumbower RD. Daily intermittent hypoxia enhances walking after chronic spinal cord injury: a randomized trial. Neurology. 2014 Jan 14;82(2):104-13. doi: 10.1212/01.WNL.0000437416.34298.43. Epub 2013 Nov 27. PMID 24285617
- See also: Neuromuscular Control & Plasticity Laboratory — http://www.rehabmed.emory.edu/pt/research/Trumbower_Lab/Homepage.html